CLINICAL TRIAL: NCT03612466
Title: A Dose Finding Study of CycloSam® (153Sm-DOTMP) Combined With External Beam Radiotherapy to Treat High Risk Osteosarcoma and Other Solid Tumors Metastatic to Bone
Brief Title: A Dose Finding Study of CycloSam® Combined With External Beam Radiotherapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdrawn before any participants could be enrolled. Issues being able to effectively recruit participants into the study.
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-8787; 7R01CA163870-06 (NIH)
Record Dates: First submitted 2018-07-30; First posted 2018-08-02 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Osteosarcoma; Bone Metastases
Keywords: dosimetry; radiopharmaceutical; radiotherapy; Maximally tolerated dose; MTD; tumor; myelosuppression
MeSH Terms: conditions — Osteosarcoma; Neoplasms | interventions — Calcium Carbonate; plerixafor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation Arm (Experimental): Dose Levels 1-3 will consist of treatment with radiopharmaceutical (153Sm-DOTMP) alone. If the maximally tolerated dose (MTD) has not been reached at Level 3, external beam radiotherapy will be added to each of Levels 4-6. Participants enrolled on Dose Levels 4-6 will be treated with external beam radiotherapy to all radiographically evident sites of disease. If an MTD has not been determined at Level 6, the study will end and Dose Level 6 will be declared the Recommended Phase 2 Dose.
  Participants will be given prophylactic / supportive treatment protocols including Calcium Carbonate, mozobil, and neupogen injectable product.
  Interventions: Drug: 153Sm-DOTMP; Radiation: External beam radiotherapy.; Drug: Calcium Carbonate; Drug: Mozobil; Drug: Neupogen Injectable Product

INTERVENTIONS:
Drug: 153Sm-DOTMP — For Levels 1- 3, the Day 1 dosages will be the same (0.5 millicurie (mCi)/kg 153Sm-DOTMP) for all levels but the Day 8 dosages will be 0.5, 1.0 and 3.0 mCi/kg respectively. For Levels 4, 5 & 6, the Day 1 dosages will be the same (0.5 mCi/kg 153Sm-DOTMP) for all levels but the Day 8 dosages will be 3, 6, then 10 mCi/kg 153Sm-DOTMP respectively.
  Other Names: CycloSam
Radiation: External beam radiotherapy. — The amount of radiation will be determined based on how much radiation was delivered to each tumor by the 153Sm-DOTMP, and will be targeted to 70 Gray (Gy)
Drug: Calcium Carbonate — Calcium carbonate will be given to participants as prophylaxis against hypocalcemia..
Drug: Mozobil — Participants who require stem cell collection will be given Mozobil to help mobilize hematopoietic stem cells into the circulation for collection.
  Other Names: plerixafor
Drug: Neupogen Injectable Product — Participants who require stem cell collection will be given Neupogen to help mobilize hematopoietic stem cells into the circulation for collection.
  Other Names: filgrastim

SUMMARY:
This is a dose finding study of a novel radiopharmaceutical agent, 153Sm-DOTMP. It will be studied alone and then in combination with external beam radiotherapy. The study design includes six cohorts, Levels 1-6. The first three cohorts of participants will receive 153Sm-DOTMP alone, and if this is determined to be safe, subsequent cohorts will receive the radiopharmaceutical followed by external beam radiotherapy.

DETAILED DESCRIPTION:
This is a dose escalation study of a new radiopharmaceutical agent, 153Sm-DOTMP. Eligible participants will have osteosarcoma metastatic to bone, other solid tumors with bone metastases, or an unresectable localized osteosarcoma. Because of anticipated prolonged myelosuppression, participants will have a peripheral blood stem cell harvest. They will then be treated with 2 doses of 153Sm-DOTMP given 7 days apart. Twenty-four days after the initial dose, stem cells will be reinfused if needed. The first three cohorts of participants will receive only radiopharmaceutical. If Dose Level 3 is not the maximally tolerated dose (MTD), subsequent dose levels will include external beam radiotherapy, administered beginning on Day 15. The dose of external beam radiotherapy will be determined by dosimetry studies performed after each administration of study agent, and will be targeted to a tumoricidal dose of radiation. All participants will have disease re-evaluation 30 days following completion of all study treatments, and then at 4, 6, 8, and 12 months, unless they experience disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor metastatic to bone, or a histologically confirmed diagnosis of osteosarcoma with either an unresectable primary tumor or metastases (including tumors with an intralesional resection).
* Measurable disease on anatomic imaging that is also avid for phosphonate compounds as demonstrated by a positive 99mTc diphosphonate bone scan.
* Adequate renal function, defined as a measured creatinine clearance >70 ml/min/1.73 m2 or normal radioisotope glomerular filtration rate (GFR).
* Adequate hematologic function, defined as a platelet count > 50,000 cells/mm3 and an absolute neutrophil count (ANC) > 500 cells/mm3
* Life expectancy of at least 8 weeks.
* Karnofsky performance status > 50%
* Subject must have adequately recovered from the effects of any prior chemotherapy, as determined by the treating physician and study team, based in part on organ function defined above. Toxicities from previous therapies must have recovered to Common Terminology Criteria for Adverse Events (CTCAE) 4.0 grade 2 or better.
* Patients must have previously received effective treatment for their underlying disease and have no potentially curative options available.

Exclusion Criteria:

* Subject has received prior radiotherapy to all known areas of current active disease or has a known contraindication to receiving radiotherapy.
* Subject is pregnant or breastfeeding.
* Patient is sexually active and does not agree to use accepted, effective forms of contraception.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Maximally Tolerated Dose | MTD will be determined based on DLTs experienced by participants during the first 42 days after administration of 153Sm-DOTMP for Dose Levels 1-3 and during the first 70 days after administration for Dose Levels 4-6
  The maximally tolerated dose (MTD) of 153Sm-DOTMP will be determined. The MTD will be defined as the dose that produces a dose limiting toxicity (DLT) in 30% of the participants. The dose limiting toxicity is the dosage at which side effects are serious enough to prevent an increase in dose or level of that treatment. DLTs will be defined as any grade 3, 4, or 5 non-hematologic toxicity experienced during a 42-70 day observation window.

SECONDARY OUTCOMES:
Overall Survival | From date of enrollment until date of death from any cause, assessed up to 60 months
  The overall survival of participants with bone metastatic osteosarcoma will be determined. Overall survival is defined as the time from enrollment in the study until death. Observation begins at study enrollment and terminates upon death of the subject.
Time To Progression | Participants will be evaluated 4, 8, and 12 months after treatment.
  The time to progression of participants with bone metastatic osteosarcoma will be determined. Time to progression is defined as the time from study enrollment until the first radiographic evidence of progressive disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST). RECIST is a set of published rules that help define whether cancer patients improve, stay the same, or get worse with treatment. This study uses the revised RECIST 1.1 guidelines.
Clinical Response Rate 30 days post treatment | 30 days post treatment
  Participants will undergo radiographic evaluation 30 days after completion of all protocol therapy. The response of each tumor to treatment will be determined based on RECIST 1.1 criteria. Clinical response will be defined as either stable disease or a decrease in the size of the tumor by radiographic imaging (which may include CT or MRI) using RECIST 1.1 criteria.
Clinical Response Rate 4 months post treatment | 4 months post treatment
  Participants will undergo radiographic evaluation 4 months after completion of all protocol therapy. The response of each tumor to treatment will be determined based on RECIST 1.1 criteria. Clinical response will be defined as either stable disease or a decrease in the size of the tumor by radiographic imaging (which may include CT or MRI) using RECIST 1.1 criteria.
Clinical Response Rate 8 months post treatment | 8 months post treatment
  Participants will undergo radiographic evaluation 8 months after completion of all protocol therapy. The response of each tumor to treatment will be determined based on RECIST 1.1 criteria. Clinical response will be defined as either stable disease or a decrease in the size of the tumor by radiographic imaging (which may include CT or MRI) using RECIST 1.1 criteria
Clinical Response Rate 12 months post treatment | 12 months post treatment
  Participants will undergo radiographic evaluation 12 months after completion of all protocol therapy. The response of each tumor to treatment will be determined based on RECIST 1.1 criteria. Clinical response will be defined as either stable disease or a decrease in the size of the tumor by radiographic imaging (which may include CT or MRI) using RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: David Loeb, MD, PhD, Principal Investigator — Children's Hospital at Montefiore
Locations (1):
- Montefiore Medical Center-Children's Hospital, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No